CLINICAL TRIAL: NCT06711653
Title: Development of Bone-vestibular Evoked Myogenic Potential
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei City Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: TCHIRB-11103021-E-F
Record Dates: First submitted 2024-11-21; First posted 2024-12-02 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2024-11

CONDITIONS: Noise; Vestibular Disorder
Keywords: bone conduction; masking; noise; random; vestibular evoked myogenic potentials
MeSH Terms: conditions — Vestibular Diseases

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Different Test Conditions (Experimental): one test group with different test conditions
  Interventions: Diagnostic Test: Vestibular evoke myogenic potential

INTERVENTIONS:
Diagnostic Test: Vestibular evoke myogenic potential — routine Vestibular test

SUMMARY:
This study aims to evaluate the effects of different masking conditions on cervical vestibular evoked myogenic potential (cVEMP) responses. Vertical-axis vibrations (VAVs) of 500-Hz short-tone bursts (STB500) and 750-Hz short-tone bursts (STB750) were used to elicit cVEMP responses. These stimuli were delivered through a Mini-Shaker placed at the vertex (Cz) under three masking conditions: no masking (NOM), speech noise masking (SNM), and random interstimulus-interval tone bursts (rISITB). The study focused on testing protocols that can potentially improve unilateral VEMP testing and explore its clinical applicability.

DETAILED DESCRIPTION:
Participants and Ethics:

The study recruited 20 healthy adults (10 males and 10 females, aged 20-37 years), all of whom had normal otoscopic findings and no history of hearing issues. Ethical approval was obtained, and all participants provided informed consent.

Bone Conduction Vibrations (BCV):

Bone-conducted vibrations were generated using a SmartEP system and delivered via a Mini-Shaker transducer. Stimuli included 500 Hz and 750 Hz short-tone bursts (STB500 and STB750), calibrated to appropriate levels, with specific rise, plateau, and fall times.

Masking Conditions:

Masking sounds included speech noise (250-1000 Hz, calibrated at 100 dB SPL) and random interstimulus-interval tone bursts (rISITB, 500 Hz, 100 dB SPL).

Testing Procedure:

Vertical-axis BCV was delivered to the vertex (Cz) while participants maintained steady neck muscle tension in specified head positions. Electrodes were placed using a standard montage for cVEMP recording. Each side was tested under three masking conditions (NOM, SNM, rISITB) with a 24-hour interval between tests. Responses were recorded bilaterally and repeated for reproducibility.

Study Focus:

The study investigates the effects of different masking conditions on response characteristics, including latencies, amplitudes, and asymmetry ratios. The aim is to refine VEMP testing protocols, explore its potential for unilateral testing, and evaluate its applicability for specific vestibular organ assessments.

ELIGIBILITY:
Inclusion Criteria:

* 20y-40y adult

Exclusion Criteria:

* Having history of hearing loss or dizziness
* failed hearing screening test
* Having history of head or neck surgery

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2022-11-07 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2023-05-01 (Actual)

PRIMARY OUTCOMES:
Vemp response rate | up to 24 weeks
  This study investigates VEMP response rates under different frequencies (500 Hz, 750 Hz) and masking conditions (no masking, speech noise, random tone bursts) to evaluate the effects of masking on VEMP responses.

CONTACTS AND LOCATIONS:
Overall Officials: Guo-She Lee, Principal Investigator — Taipei City Hospital
Locations (1):
- Taipei City Hospital, Taipei, Taiwan